CLINICAL TRIAL: NCT03448874
Title: Seal-G MIST System Safety Study [SEALAR Study]
Brief Title: Seal-G MIST (Minimally Invasive Sealant/Spray Technology) System Safety Study [SEALAR Study]
Acronym: SEALAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company will design a new study
Sponsor: Sealantis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLG-072-06
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer; Diverticulitis Colon
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis, Colonic

STUDY DESIGN:
Intervention Model Description: Controlled, Randomized, single blind study
Who Masked: Participant
Masking Description: This study is single blinded. The subject will be blinded to the treatment arm; however, by nature of the type of the proposed study, blinding of the investigator/ surgeon is not feasible. In order to minimize bias, subjects will be randomized during the surgery upon confirmation of the intra-operative exclusion criteria. This will ensure that the surgeon will not know prior to surgery and until completion of anastomosis creation, whether or not Seal-G MIST will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seal-G MIST System (Experimental): Seal-G MIST System is a surgical sealant that will be applied adjunctively to standard closure techniques for reinforcement and protection of gastrointestinal anastomoses.
  Interventions: Device: Seal-G MIST System
- Standard of care (No Intervention): Patients in the control arm will receive the standard of care [SOC] for colorectal resection surgery with primary anastomosis (no additional intervention)

INTERVENTIONS:
Device: Seal-G MIST System — Seal-G MIST is an adjunct device that will be applied adjunctively to cover standard closure techniques.
  Other Names: Seal-G MIST
  Arms: Seal-G MIST System

SUMMARY:
The purpose of this study is to evaluate safety of Seal-G MIST System in reinforcing colorectal anastomosis, in subjects undergoing colorectal surgery.

DETAILED DESCRIPTION:
Study procedures:

Pre-surgery:

* Screening will be performed among adult subjects who are scheduled for an elective colorectal surgery. Once potential eligibility to the study is determined based on the study's inclusion/exclusion criteria, study procedures will be explained to the candidate and participation will be offered.
* Informed consent process.
* Pre-surgery assessments will be according to the routine practice at the site and determined by the treating physician.

Intra-operative:

* During the surgery, after confirmation of the intra-operative exclusion criteria, completion of anastomosis creation and only after leak test was performed , subjects will be allocated to one of the two treatment arms with a 1:1 ratio based on a randomization scheme (either to the Standard of care (SOC) or to Seal-G MIST arms).
* Device (Seal-G MIST System) application (to Seal-G MIST treatment arm only).

Post-operative follow-up:

* Subjects will be followed during post-operative period until discharge from the hospital for clinical and subclinical leaks according to the SOC.
* In an event of suspected anastomotic leak, patient will be treated according to severity of leak and PI clinical judgement (conservative treatment, drainage, diversion, anastomosis take down).
* Subjects will be followed up for leaks and related AE/SAEs at the day of the surgery and for a period of 15 weeks (±2 weeks) post-surgery, including the following activities:

  * Daily while hospitalized (in accordance with the site routine procedures)
  * At 1 month (±1 week) and 15 weeks (±2 weeks) post-surgery (Hospitalization for elective procedure (i.e. chemotherapy treatments) will not be considered as SAEs)

ELIGIBILITY:
Inclusion Criteria:

1. Subject >18 years
2. Subject is scheduled for elective open or laparoscopic colorectal resection (including left colectomy, sigmoidectomy, anterior resection, subtotal colectomy) surgery (including robotic) involving the creation of circular stapler anastomosis
3. Subject signs and dates a written Informed Consent Form, indicates an understanding of the study procedures and follow-up requirements and is willing to comply with them

Exclusion Criteria:

1. Anastomosis is expected to be ≤ 10cm from anal verge
2. Surgery involves stoma creation
3. Subject who underwent a prior pelvic radiation therapy
4. Subject with a BMI > 40 or <19
5. Subject with American Society of Anesthesiologists (ASA) status higher than 3
6. Albumin level < 3 gr/dl
7. Hemoglobin level < 8 g/dl on day of surgery
8. Subject has a diagnosis of bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, and carcinomatosis
9. Subject treated with immunosuppressive agents within 28 days prior to study enrollment (including corticosteroids)
10. Serious or uncontrolled co-existent diseases (e.g. severe cardiovascular disease, congestive heart failure, recent myocardial infarction within 6 months from surgery, significant vascular disease, active or uncontrolled autoimmune disease, active or uncontrolled infection, uncontrolled diabetes mellitus with episodes of hospitalization due to hypo or hyperglycemia within 6 months of surgery)
11. Subject known to have distant metastases, such as liver, lung, bone etc. metastases (not including local and regional lymph nodes)
12. Subject with known sensitivity to Indigo carmine dye (E132)
13. Subject who according to the investigator clinical judgement is not suitable for participation in the study
14. Subject with a life expectancy of less than 1 year
15. Subject requires more than one anastomosis during the surgery
16. Subject is scheduled for another surgery during the follow up period of this study
17. Subject participating in any other study involving an investigational (unapproved) drug or device
18. Woman who is known to be pregnant or breast-feeding or woman who is planning pregnancy or breast-feeding in the 5 next months
19. Vulnerable subjects (e.g. mentally handicapped, prisoners, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of overall subject pre-specified* procedure related Adverse Events | up to 15 weeks (±2 weeks) post-surgery
  Pre-specified procedure related Adverse Event: Wound infection; Bowel obstruction and Post-operative ileus; Anastomotic stricture; Anastomotic leak; Collection/Abscess; Urinary retention/Urinary Tract Infection; Renal failure; Hepatic failure; Peritoneal metastasis; Staple-line bleeding; Allergic reaction; Re-intervention (Including but not limited to re-operation; stoma).

SECONDARY OUTCOMES:
Incidence of clinical anastomotic leaks | up to 15 weeks (±2 weeks) post-surgery
  Anastomotic leak (AL) is defined as evidence of a defect in the intestinal wall integrity at the anastomotic site leading to local or general peritonitis, abscesses in the proximity of the anastomosis and/or fistula, fecal or purulent discharge from drains.
Incidence of subclinical/ radiological leaks | up to 15 weeks (±2 weeks) post-surgery
  As assessed from Adverse event/Serious Adverse Event reporting form
Incidence of Serious Adverse Events (SAE) complications | up to 15 weeks (±2 weeks) post-surgery
  According to Serious Adverse Event (SAE) definition from Medical Device Directive (MEDDEV 2.7/3, Rev 3, May 2015)
Incidence of collection/abscess without demonstrated leak | up to 15 weeks (±2 weeks) post-surgery
  According to Adverse event reporting form
Incidence of reoperation | up to 30 days post-surgery
  According to Adverse event/Serious Adverse Event reporting form
Incidence of postoperative mortality | up to 15 weeks (±2 weeks)
Hospital length of stay | From date of surgery until the time for "Ready to be discharged" (in days), an average of 10±4 days
Incidence of "deployment failure" | during surgery
  only for treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Kamar, MD, Study Director — Chief Medical Officer

IPD SHARING:
Plan to Share IPD: Undecided